CLINICAL TRIAL: NCT05354011
Title: Effects of Kinesiotaping With and Without Active Release Technique on Pain, Grip Strength, Functional Disability and Range of Motion in Patients With Carpal Tunnel Syndrome
Brief Title: Effects of Kinesiotaping With and Without Active Release Technique in Patients With Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0111 Janisar
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: CTS; Wrist pain; Disability; Kinesiotaping; Active Release Technique
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Athletic Tape

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping (Experimental): Kinesiotape will be applied toward the start of the week, to remain on for 5 days with a multi day rest for an aggregate of about a month.
  Interventions: Other: Kinesiotape
- Active Release Technique (Experimental): kinesiotaping and active release technique will be applied 3 times a week for 2 week
  Interventions: Other: Active Release Technique

INTERVENTIONS:
Other: Kinesiotape — Tape with a width of 5 cm and a thickness of 0.5 mm will be utilized. Kinesio Tex I Strip is estimated from elbow to fingertips and cut. It will be collapsed roughly two squares from the end and cut into two triangles on the overlay. The third and fourth fingers are fallen through openings and Kinesio Tex is applied on the dorsum of the hand with no strain. The situation of elbow extension, wrist extension, and radial deviation is given, and Kinesio Tex will be applied from hand to medial epicondyle with 15%-25% tension and end at medial epicondyle with no strain
  Arms: Kinesiotaping
Other: Active Release Technique — This group will receive Kinesiotaping with the same method along with Active release technique will be performed on group 2. We will apply profound tension at the region of tenderness while the patient is told to effectively move the injury site from a shortened to lengthened position. The setting of a contact point close to the injury and making the patient move in a way that creates a longitudinal sliding movement of delicate tissues e.g. nerves, ligaments and muscles underneath the contact point.
  Arms: Active Release Technique

SUMMARY:
The goal of this study is to compare the effects of Kinesiotaping and Active Release Technique in patients with CTS to see which method is better for improving Pain, Grip Strength, Range of Motion and functional disability.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a common nerve entrapment condition that causes pain, numbness, tingling and weakness in the hand and wrist. People suffering from CTS complain of pain, decreased ROM, loss of grip strength and in severe cases, disability. This happens when there is an increased pressure within the wrist on a nerve called "Median Nerve". This nerve provides sensations to the thumb, index, middle and half of the ring finger. People who are most susceptible to CTS are computer/keyboard workers. High force, extreme wrist motions, vibrations are causes. Other factors like genetics and pregnancy can also cause CTS. There are a lot of treatment options for CTS such as use of orthotics, steroidal injections, surgery and physical therapy. The aim of this study will be to determine the effects of kinesiotaping with and without active release technique on pain, grip strength, functional disability and range of motion in patients with carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients having symptoms for less than 1 year.

  * Age above 18 years.
  * Patients having positive Tinel and Phalen test.
  * Pain in the median nerve distribution with minimum score of 3 on NPRS. Ability to read and understand the study instructions and written consent form

Exclusion Criteria:

* Having any secondary entrapment neuropathy like diabetes, inflammatory arthritis, and hypothyroidism.

  * Pregnancy Skin infection on the forearm, cervical radiculopathy or polyneuropathy.
  * Previous history of Carpal Tunnel Decompression Surgery.
  * Corticosteroid injection into the Carpal Tunnel.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
NPRS | 3 months
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain)
hand dynamometer | 3 months
  A hand dynamometer is an evaluation tool that's used to measure isometric grip force (hand grip strength). Some versions use hydraulics to measure the force while others use electronic load cells. Once the grip position is adjusted, the user holds the handle and squeezes the handle
Boston CTS Questionnaire | 3 months
  The Boston Carpal Tunnel Questionnaire (BCTQ) is a disease-specific measure of selfreported symptom severity and functional status. It is frequently used in the reporting of outcomes from trials into interventions for carpal tunnel syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Nosheen Manzoor, MS, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zainab J, Manzoor N, Bashir MS, Noor R, Ikram M. Effects of kinesio taping with and without active release technique in carpal tunnel syndrome. Hand Surg Rehabil. 2024 Feb;43(1):101633. doi: 10.1016/j.hansur.2024.101633. Epub 2024 Jan 6. PMID 38190964